CLINICAL TRIAL: NCT05625958
Title: Multicentre, Non-randomised Clinical Study Evaluating the Safety and Efficacy of a Cilioscleral Interposition Device ("CID") v2.2 in Glaucoma Surgery
Brief Title: Clinical Study Evaluating the Efficacy and Safety of CID v2.2 in Glaucoma Surgery
Acronym: SAFARI4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciliatech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAFARI 4
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma, Open-Angle; Glaucoma, Narrow Angle
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Angle-Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cilioscleral Interposition Device (Experimental): Any patients corresponding to inclusion / exclusion criteria
  Interventions: Device: Cilioscleral Interposition Device

INTERVENTIONS:
Device: Cilioscleral Interposition Device — Surgical placement of SV22 cilioscleral interposition device in the supraciliary space

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of implanting a new version of an interposition supraciliary implant (SV22) as a stand-alone therapy for lowering intraocular pressure (IOP) in patients with primary open and narrow angle glaucoma who have failed at least one class of topical medical therapy

DETAILED DESCRIPTION:
29 patients will be included in this 36 months interventional study.

All patients shall be indicated for glaucoma surgery alone (not combined with cataract), and will undergo incisional glaucoma therapy, including a simplified surgical technique allowing the placement of an interposition supraciliary permanent device.

Several patient data like safety events, IOP, visual capacity or associated pharmacological treatments will be recorded pre and post-operatively all along the follow-up.

Purpose is to ensure device safety, and verify IOP and associated pharmacological treatment reduction after surgery, and evolution along follow-up.

ELIGIBILITY:
Inclusion Criteria To be included in the study, all patients must meet all the following inclusion criteria:

Patient:

1. 18 years or older
2. Able to understand study requirements
3. Able and willing:

   1. To provide written consent on the EC-approved Informed Consent Form,
   2. To comply with all study requirements, including required study follow-up visits' agenda

   Eye:
4. Glaucoma (angle from 1 to 4 according to Schaffer grade), including pseudo exfoliative and pigmentary glaucoma, which meets the following:

   1. Vertical C/D ratio on fundoscopic exam ≤ 0.9, or OCT demonstrating a thinness of the nerve fibre layer at the p<5% level as defined by the instrument's built-in age-adjusted normative database,
   2. Glaucoma visual field with -15 < MD < 0dB (Humphrey) or 0 < MD < 15 dB (Octopus)
5. Pharmacological treatments: glaucoma not adequately controlled by 1 to 3 different IOP-lowering medication(s), given each for at least one month prior to Screening,
6. IOP:

   1. if using 1 or 2 IOP-lowering medications, IOP is between 18 mmHg and 30 mmHg in the study eye at Screening visit
   2. if using 3 IOP-lowering medications, IOP is between 18 mmHg and 25 mmHg in the study eye at Screening visit
7. Having the indication for glaucoma surgery alone (no concomitant cataract surgery)
8. Central Corneal Thickness between 480 to 620 µm
9. Gonioscopy confirming normal angle anatomy at site of implantation. Angle anatomy may include Peripheral Anterior Synechiae (PAS) of up to maximum of 3 clock hours if not present parallel to the proposed site of device implantation.

Exclusion criteria Patients will not participate in this clinical study if they meet any of the following criteria:

Patient:

1. Patient with a known allergy to any of the constituents of the products used in this study or known steroid responder
2. Patient already included in another study
3. A person protected by law (temporary or permanent guardianship) or not capable of discernment
4. Patient who may not assist to all follow-up visits (because of frequent travelling, or living in remote area, or limited moving capacities, …)
5. Pregnant or nursing woman at the date of inclusion (only for women of childbearing potential: positive urine pregnancy test at screening)
6. With uncontrolled systemic disease that, in the opinion of the Investigator, would put the subject's health at risk and/or prevent the subject from completing all study visits (e.g. inability to reliably complete visual field testing over the course of the study, or take glaucoma medications (e.g. Parkinson's disease), or uncontrolled systemic disease (diabetes, hypertension) that could compromise participation in the study, …)
7. Who have a new or modified prescription for a systemic treatment that could influence IOP within one month prior to inclusion, or who are aware of a future change in their systemic treatment, or if their medical condition indicates that their systemic treatment may change in the future
8. Chemotherapy in the last 6 months before surgery

   Eye:
9. Inflammatory, congenital, malignant, traumatic, uveitic, neovascular glaucoma or iridocorneal endothelial syndrome (ICE syndrome)
10. Fast progressing or very severe glaucoma or any condition requiring a filtering surgery
11. History of any incisional glaucoma surgery or implantable glaucoma device
12. Prior SLT, ALT or MLT
13. Eye surgery (other than glaucoma) less than 6 months ago, or presenting sequelae of previous eye surgery or trauma
14. Eye with uncontrolled IOP despite 4 IOP-lowering medications prescribed for more than a month
15. Eye with severe OSD and / or severe dry eye defined as Oxford score ≥ 4
16. Inability to obtain accurate IOP measurement throughout the study (e.g. history of corneal surgery, corneal opacities or disease/pathology)
17. Conditions associated with elevated episcleral venous pressure such as active thyroid orbitopathy, cavernous sinus fistula, Sturge Weber syndrome, orbital tumors, orbital congestive disease
18. Any known ocular condition that may require intraocular intervention during the protocol required follow-up period
19. Premature or mature cataract (initial cataract are accepted)
20. Any condition that prevents the investigational device implantation in the superior and nasal region of the eye
21. Pre-existing ocular or systemic pathology that may, in the opinion of the Investigator, cause post-operative complications
22. Non laser retinal surgery
23. Previous cyclodestructive or scleral buckling procedure
24. History of complicated cataract surgery (as posterior capsular rupture, vitreous loss)
25. History of silicone oil
26. Ocular steroid in the planned study eye or systemic steroid use in the last 3 months before surgery
27. Use of oral hypotensive glaucoma medications for treatment of the fellow eye
28. Axial length <20 mm
29. Severe myopia defined as spherical correction < -8 Diopters
30. Best corrected distant visual acuity of 0.1 (20/200) or worse in the study or fellow eye
31. Peripheral synechia at the angle
32. Closed angle
33. Peripheral laser iridotomy in the last 7 days before planned surgery
34. Epithelial or fibrous downgrowth
35. Any kind of endothelial dystrophy
36. Severe blepharitis
37. Chronic or recurrent uveitis
38. Conjunctiva showing keratitis, fine conjunctiva, erosion or abnormal vascularisation
39. Active iris neovascularization, rubeosis, proliferative retinopathy, diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders), vitreous haemorrhage, preretinal haemorrhage, choroidopathy or other ophthalmic disease that could confound study results
40. Scleral fixation IOL
41. Lens dislocation or subluxation
42. Vitreous loss in the anterior chamber

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Assess post-op IOP reduction | 6 months
  Mean change in medicated IOP and IOP-lowering pharmacological treatments from baseline and 6 months after surgery

SECONDARY OUTCOMES:
Change in medicated IOP and IOP-lowering treatments | baseline and 12, 24, and 26 months after surgery
  Mean change in medicated IOP and IOP-lowering pharmacological treatments
Decrease in IOP from baseline up to 36 months post-operatively | baseline up to 6, 12, 24, and 36 months post-operatively
  Proportion of eyes with greater than or equal to 20% decrease in IOP from baseline up to 36 months post-operatively with IOP lowering medication
Mean medicated IOP | baseline, 6, 12, 24, and 36 months after surgery
  Mean medicated IOP at baseline and up to 36 months after surgery
Mean number of IOP lowering treatments | baseline, 6, 12, 24, and 36 months after surgery
  Mean number of IOP lowering pharmacological treatments at baseline and up to 36 months after surgery
Absolute success rate: proportion of med-free eyes | 6, 12, 24, and 36 months
  Proportion of med-free eyes with IOP decrease of greater than or equal to 20% from baseline and below 18 mmHg up to 36 months after surgery
Qualified success rate: proportion of eyes with IOP decrease | 6, 12, 24, 36 months
  Proportion of eyes with IOP decrease of greater than or equal to 20% from baseline and below 18 mmHg up to 36 months after surgery
Rate of patients with reduction of IOP at each visit | 36 months
  Rate of patients with at least a 20%, 30%, 40% and more than 50% reduction in IOP at each visit vs baseline, with and without IOP lowering pharmacological treatments
Proportion of eyes free of ocular hypertensives | 6, 12, 24, and 36 months after surgery
  Proportion of eyes free of ocular hypotensive medications at 6, 12, 24 and 36 months after surgery
Proportion of eyes with IOP between 6 and 18 mmHg with and without IOP lowering treatments | 6, 12, 24 and 36 months after surgery
  Proportion of eyes with IOP ≥6 mmHg and ≤ 18 mmHg, with and without IOP-lowering pharmacological treatments at 6, 12, 24 and 36 months after surgery
Proportion of eyes with IOP between 6 and 16 mmHg with and without IOP lowering treatments | 6, 12, 24 and 36 months after surgery
  Proportion of eyes with IOP ≥6 mmHg and ≤ 16 mmHg, with and without IOP-lowering pharmacological treatments at 6, 12, 24 and 36 months after surgery
Number of adjunctive therapies | 36 months
  Average number of adjunctive therapies (needling, goniopuncture, SLT,
  …) performed up to 36 months postoperatively
Patient rate without filtering bleb | 6, 12, 24 and 36 months after surgery
  Rate of patients without filtering bleb, average duration of filtering blebs at 6, 12, 24 and 36 months after surgery
Surgical implantation evaluation | 1 day
  To evaluate the surgical procedure (duration of operation, ease of implantation)
Assess patient experience post-operatively | 1 and 7 days, then at 1, 6, 12, 24 and 36 months after surgery
  To describe patient experience following surgery using questions asked by the surgeon, for pain (Yes/No), quality of vision (deteriorated, stable, improved) and sensation in the eye (discomfort / nothing to declare) at 1 and 7 days, then at 1, 6, 12, 24 and 36 months after surgery
Describe patient satisfaction post-operatively | 1, 6, 12, 24 and 36 months after surgery
  To describe patient satisfaction following surgery using questionnaires (VAS scale) for comfort and satisfaction at 1, 6, 12, 24 and 36 months after surgery
Assess patient quality of life | 1, 6, 12, 24 and 36 months after surgery
  To describe changes in quality of life using EQ5D-5L questionnaire at 1, 6, 12, 24 and 36 months after surgery
Rate of device related ocular adverse events and adverse device effects | up to 36 months
  Rate of intraoperative and post-operative device related ocular adverse events and adverse device effects
Safety examination findings | up to 36 months
  Slit lamp, gonioscopy and fundus findings
Rate of Best Corrected Visual Acuity | 6, 12, 24 and 36 months after surgery
  Rate of Best Corrected Visual Acuity variation (BCVA) at 6, 12, 24 and 36 months after surgery
Rate of Visual Field Mean Deviation variation | 6, 12, 24 and 36 months after surgery
  Rate of Visual Field Mean Deviation variation (VF MD) at 6, 12, 24 and 36 months after surgery
Rate of C/D ratio mean deviation | 6, 12, 24 and 36 months after surgery
  Rate of C/D ratio mean deviation at 6, 12, 24 and 36 months after surgery
Rate of sight threatening events | up to 36 months
  Rate of sight threatening events
Rate of change in endothelial cell density (ECD) and central corneal thickness (CCT) | 6, 12, 24 and 36 months after surgery
  Rate of change in endothelial cell density (ECD) and central corneal thickness (CCT) at 6, 12, 24 and 36 months after surgery
Rate of occurrence of SUPRAFLOW V2.2 movements | 6, 12, 24 and 36 months after surgery
  Rate of occurrence of SUPRAFLOW V2.2 movements inside the supraciliary space at 6, 12, 24 and 36 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Julian GARCIA FEIJOO, Pr, Principal Investigator — Clinica San Carlos
Locations (6):
- Spain (6):
  - Hospital Clínic of Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos. Servicio de Oftalmología, Madrid
  - OMIQ Research, Sabadell
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet. Servicio de Oftalmología., Zaragoza

IPD SHARING:
Plan to Share IPD: No